CLINICAL TRIAL: NCT01341457
Title: A Phase 1 Dose-Escalation Study of LY2603618 in Combination With Gemcitabine in Japanese Patients With Solid Tumors
Brief Title: A Study of LY2603618 in Combination With Gemcitabine in Participants With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13574; I2I-JE-JMME (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-04-19; First posted 2011-04-25 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Solid Tumors
MeSH Terms: interventions — LY2603618; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2603618 + Gemcitabine (Experimental): Gemcitabine 1000 milligrams per meter squared (mg/m^2) administered intravenously on days 1, 8 and 15 of at least one 28-day cycle. 170 or 230 mg LY2603618 administered intravenously on days 2, 9 and 16 of at least one 28-day cycle.
  Participants experiencing benefit may continue on the combination therapy until discontinuation criteria are met.
  Interventions: Drug: LY2603618; Drug: Gemcitabine

INTERVENTIONS:
Drug: LY2603618 — Administered intravenously
Drug: Gemcitabine — Administered intravenously
  Other Names: LY188011

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of LY2603618 in combination with the standard dose of gemcitabine up to the global recommended dose of LY2603618 in Japanese participants with solid advanced or metastatic tumors.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological or imaging evidence of a diagnosis of cancer that is advanced and/or metastatic disease
* Participant who is planned to have gemcitabine therapy at the proposed doses because he/she was not able to benefit from standard therapy and/or therapies known to provide clinical benefit or there is no standard therapy for the advanced and/or metastatic disease globally
* Have given written informed consent prior to any study-specific procedures
* Have adequate hematologic, hepatic and renal function
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous therapies for cancer, including chemotherapy, cancer-related hormonal therapy, or other investigational therapy for at least 30 days (42 days for mitomycin C or nitrosoureas) prior to study enrollment and recovered from the acute effects of therapy
* Prior radiation therapy for treatment of cancer is allowed to less than 25% of the bone marrow, and participants must have recovered from the acute toxic effects of their treatment prior to study enrollment. Prior radiation to the whole pelvis is not allowed. Prior radiotherapy must be completed at least 30 days prior to study enrollment
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the study and for 3 months after the last infusion of study drug
* Females with child bearing potential (not surgically sterilized and between menarche and 1 year post menopause) must have had a negative urine pregnancy test less than 7 days prior to the enrollment
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have an estimated life expectancy of at least 12 weeks

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical study involving an off-label use of an investigational drug or device (other than the study drug used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have serious preexisting medical conditions or serious concomitant systemic disorders that would compromise the safety of the participant or his/her ability to complete the study
* Have interstitial pneumonitis or pulmonary fibrosis, or previous history of them
* Have symptomatic central nervous system malignancy or metastasis
* Have current active infection
* Females who are pregnant or lactating
* Have known positive test results in human immunodeficiency virus (HIV), hepatitis B surface antigen (HBSAg), or hepatitis C antibodies (HCAb)
* Participants with acute or chronic leukemia or with any other disease likely to have a significant bone marrow infiltration
* Have previously completed or withdrawn from this study or any other study investigating LY2603618 or any other checkpoint kinase (Chk1) inhibitor
* Have known allergy to gemcitabine or LY2603618 or any ingredient of gemcitabine or LY2603618 (like Captisol®)
* Have an abnormal electrocardiogram (ECG) result that would put the participant at unnecessary risk in the opinion of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant study completion is defined as a participant completing the primary and secondary objective assessments.
Groups:
- 170 mg LY2603618 + Gemcitabine: Gemcitabine 1000 milligrams per meter squared (mg/m²) administered intravenously (IV) on days 1, 8 and 15 of at least one 28-day cycle. 170 mg LY2603628 administered IV on days 2, 9 and 16 of at least one 28-day cycle.
  Participants experiencing benefit may continue on the combination therapy until discontinuation criteria are met.
- 230 mg LY2603618 + Gemcitabine: Gemcitabine 1000 mg/m² administered IV on days 1, 8 and 15 of at least one 28-day cycle. 230 mg LY2603628 administered IV on days 2, 9 and 16 of at least one 28-day cycle.
  Participants experiencing benefit may continue on the combination therapy until discontinuation criteria are met.
Period: Overall Study
Arm/Group | 170 mg LY2603618 + Gemcitabine | 230 mg LY2603618 + Gemcitabine
Started | 7 | 10
Received at Least One Dose of Study Drug | 7 | 10
Completed | 5 | 10
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 170 mg LY2603618 + Gemcitabine | 230 mg LY2603618 + Gemcitabine | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.33) | 60.8 (6.81) | 61.3 (7.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 1 | 9 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 10 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLT is defined as adverse event (AE) during Cycle 1 (Days 1 through 28) that was possibly related to the study drug and toxicities considered by the investigator as dose limiting. A summary of other nonserious AEs, and all serious adverse events (SAE's), regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Cycle 1 (28 Days)
Population: Participants who completed the first cycle of study treatment or who discontinued study treatment due to a DLT. There was one participant in the 170 mg LY2603618 treatment group that had an insufficient number of doses of gemcitabine to evaluate DLT.
Measure: Count of Participants; unit: Participants
Groups:
- 170 mg LY2603618 + Gemcitabine: Gemcitabine 1000 mg/m² administered IV on days 1, 8 and 15 of at least one 28-day cycle. 170 mg LY2603628 administered IV on days 2, 9 and 16 of at least one 28-day cycle.
  Participants experiencing benefit may continue on the combination therapy until discontinuation criteria are met.
Arm/Group | 170 mg LY2603618 + Gemcitabine | 230 mg LY2603618 + Gemcitabine
Number analyzed (Participants) | 6 | 10
Participants | 1 | 2

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) of LY2603618
Time Frame: Cycle 1 (days 2 and 16) & 2 (day 2): Predose, End of Infusion, 1 hour (h), 3h, 6h, 24h (days 3 and 17), 48h (days 4 and 18 cycle 1 only), 72h (days 5 and 19)
Population: All randomized participants who received at least one dose of study drug and have had PK samples collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per Milliliter (ng/mL)
Arm/Group | 170 mg LY2603618 + Gemcitabine | 230 mg LY2603618 + Gemcitabine
Number analyzed (Participants) | 7 | 10
Nanograms per Milliliter (ng/mL)
  Cycle 1 Day 2 | 3610 (37) | 3920 (56)
  Cycle 1 Day 16: number analyzed (Participants) | 5 | 7
  Cycle 1 Day 16 | 3510 (41) | 4120 (42)
  Cycle 2 Day 2: number analyzed (Participants) | 4 | 8
  Cycle 2 Day 2 | 3290 (24) | 3570 (38)

3. Secondary Outcome: Number of Participants With Best Overall Response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) (Best Overall Response)
Description: Participants achieved disease control if they had a best overall response of PR, CR or SD according to RECIST v1.1 (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD); PR at least 30% decrease and PD at least 20% increase in the sum of diameter of target lesions; CR: disappearance of all target lesions). Two determinations of PR or better before progression, but not qualifying for a CR, are required for a best response of PR. Best response of SD is defined as disease that does not meet the criteria for CR, PR or PD and has been evaluated at least 6 weeks after the first gemcitabine administration.
Time Frame: Baseline to Measured Progressive Disease (Up to 52 Months)
Population: All randomized participants who received at least one dose of study drug and had measurable lesion(s).
Measure: Number; unit: participants
Arm/Group | 170 mg LY2603618 + Gemcitabine | 230 mg LY2603618 + Gemcitabine
Number analyzed (Participants) | 7 | 10
participants | 2 | 5

4. Secondary Outcome: PK: Area Under the Plasma Concentration vs. Time Curve From Time Zero to Infinity [AUC(0-∞)] of LY2603618
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of study drug and have had PK samples collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | 170 mg LY2603618 + Gemcitabine | 230 mg LY2603618 + Gemcitabine
Number analyzed (Participants) | 7 | 10
nanograms*hour per milliliter (ng*h/mL)
  Cycle 1 Day 1 | 43900 (74) | 37200 (71)
  Cycle 1 Day 16: number analyzed (Participants) | 5 | 7
  Cycle 1 Day 16 | 52600 (91) | 39000 (40)
  Cycle 2 Day 2: number analyzed (Participants) | 4 | 8
  Cycle 2 Day 2 | 47800 (59) | 35800 (33)

5. Secondary Outcome: PK: Cmax of Gemcitabine
Time Frame: Cycle 1 (days 1 and 15) & 2 (day 1): Predose, End of Infusion, 10 minutes (m), 30m, 60m, 120m
Population: All randomized participants who received at least one dose of study drug and have had PK samples collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- LY2603618 + Gemcitabine: Gemcitabine 1000 milligrams per meter squared (mg/m²) administered intravenously (IV) on days 1, 8 and 15 of at least one 28-day cycle. 170 or 230 mg LY2603628 administered IV on days 2, 9 and 16 of at least one 28-day cycle.
  Participants experiencing benefit may continue on the combination therapy until discontinuation criteria are met.
Arm/Group | LY2603618 + Gemcitabine
Number analyzed (Participants) | 17
ng/mL
  Cycle 1 Day 1 | 23000 (16)
  Cycle 1 Day 15: number analyzed (Participants) | 12
  Cycle 1 Day 15 | 24700 (25)
  Cycle 2 Day 1: number analyzed (Participants) | 12
  Cycle 2 Day 1 | 18100 (27)

6. Secondary Outcome: PK: Cmax of Gemcitabine Metabolite Deoxydifluorouridine (dFdU)
Time Frame: Cycle 1 (days 1 and 15) & 2 (day 1): Predose, End of Infusion, 10 minutes (m), 30m, 60m, 120m
Population: All randomized participants who received at least one dose of study drug and have had PK samples collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LY2603618 + Gemcitabine
Number analyzed (Participants) | 17
ng/mL
  Cycle 1 Day 1 | 40100 (15)
  Cycle 1 Day 15: number analyzed (Participants) | 12
  Cycle 1 Day 15 | 38600 (18)
  Cycle 2 Day 1: number analyzed (Participants) | 12
  Cycle 2 Day 1 | 38400 (18)

7. Secondary Outcome: PK: AUC(0-∞) of Gemcitabine
Time Frame: Cycle 1 (days 1 and 15) & 2 (day 1): Predose, End of Infusion, 10 minutes (m), 30m, 60m, 120m
Population: All randomized participants who received at least one dose of study drug and have had PK samples collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | LY2603618 + Gemcitabine
Number analyzed (Participants) | 17
ng*h/mL
  Cycle 1 Day 1 | 11600 (17)
  Cycle 1 Day 15: number analyzed (Participants) | 12
  Cycle 1 Day 15 | 12300 (32)
  Cycle 2 Day 1: number analyzed (Participants) | 12
  Cycle 2 Day 1 | 9530 (23)

8. Secondary Outcome: PK: AUC(0-∞) of Gemcitabine Metabolite dFdU
Time Frame: Cycle 1 (days 1 and 15) & 2 (day 1): Predose, End of Infusion, 10 minutes (m), 30m, 60m, 120m
Population: All randomized participants who received at least one dose of study drug and have had PK samples collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | LY2603618 + Gemcitabine
Number analyzed (Participants) | 17
ng*h/mL
  Cycle 1 Day 1: number analyzed (Participants) | 16
  Cycle 1 Day 1 | 126000 (28)
  Cycle 1 Day 15: number analyzed (Participants) | 10
  Cycle 1 Day 15 | 136000 (32)
  Cycle 2 Day 1: number analyzed (Participants) | 11
  Cycle 2 Day 1 | 142000 (23)

ADVERSE EVENTS:
Arm/Group | 170 mg LY2603618 + Gemcitabine | 230 mg LY2603618 + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 0/7 | 2/10
Other Adverse Events (participants affected / at risk) | 7/7 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 170 mg LY2603618 + Gemcitabine (N=7) | 230 mg LY2603618 + Gemcitabine (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 170 mg LY2603618 + Gemcitabine (N=7) | 230 mg LY2603618 + Gemcitabine (N=10)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (10)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 5 (6) | 8 (18)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (4)
Fatigue (General disorders) | 2 (3) | 6 (9)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (5) | 4 (11)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 4 (5)
Amylase increased (Investigations) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (6)
Blood alkaline phosphatase increased (Investigations) | 2 (3) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (3) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
Blood magnesium increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 3 (3)
Haemoglobin decreased (Investigations) | 7 (8) | 8 (8)
Neutrophil count decreased (Investigations) | 5 (15) | 9 (85)
Platelet count decreased (Investigations) | 7 (9) | 6 (47)
White blood cell count decreased (Investigations) | 6 (19) | 9 (84)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (6) | 6 (14)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin striae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (4) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days